CLINICAL TRIAL: NCT04770727
Title: Feasibility of a Group Intervention Using Cognitive Behavioural Therapy (CBT) to Reduce Anxiety for Children Aged 12-17 With Food Allergy.
Brief Title: CBT Group Intervention for Children With Food Allergy and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHMS 20-21 002 EGA
Record Dates: First submitted 2021-02-18; First posted 2021-02-25 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Food Allergy in Children
Keywords: Food Allergy; Anxiety; Young People
MeSH Terms: conditions — Food Hypersensitivity; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workshop Intervention (Experimental): A psychoeducation workshop will be provided alongside a workbook containing the content to review and refresh skills learnt. The psychoeducational intervention will be delivered by trainee clinical psychologists with interests in food allergy and delivered in line with a protocol.
  Interventions: Behavioral: CBT workshop
- Treatment as usual (No Intervention): Adolescents randomised to the control arm will continue treatment as usual and receive the workshop materials after the active treatment group have completed their final follow-up at 3 months.

INTERVENTIONS:
Behavioral: CBT workshop — The CBT based intervention for adolescents will include psychoeducation on food allergy and anxiety and also focus on providing skills, knowledge and support.
  Arms: Workshop Intervention

SUMMARY:
The research will design and evaluate a CBT based intervention to support children aged 11-17 with food allergies. The research on this population has shown that they can experience high levels of anxiety in management of their allergy which can have a significant impact on quality of life. However, the research exploring psychological interventions is limited. CBT has a wide evidence base from NHS settings delivering interventions to support those with various health conditions. In addition, CBT has been shown to be effective for supporting adolescents manage their health-related anxiety. The investigators are interested in the feasibility of designing and implementing a one day workshop aimed at adolescents with food allergy and self-reported anxiety. The group workshop will involve psychoeducation on anxiety, skills and techniques to manage anxiety, relaxation and how to set goals in relation to their food allergy. It will involve 2 'arms', one where participants will attend the group and the other 'control arm' where they will not attend the group but they will receive materials from the group once the evaluation is complete. All participants will be asked to complete questionnaires that measure level of anxiety, food allergy quality of life and coping skills at baseline, time of workshop, one month follow up and three month follow up. There will also be an opportunity for participants to volunteer to take part in a follow up interview to evaluate the workshop and also to contribute more to the research on what this population requires in terms of a psychological intervention.

DETAILED DESCRIPTION:
Food allergy is an increasing public health concern, with Westernised countries reporting prevalence of diagnosed allergies of up to 10%, most notably among younger children. Over the last few decades, the number of people diagnosed with food allergy has been increasing, as has the awareness of the psychological burden of living with a food allergy. As the symptoms lie on a spectrum with fatal anaphylaxis being a possible result of exposure, avoidance of the allergen and having access to emergency medication (e.g. adrenaline auto-injectors) remains the primary care for management Unlike other allergies which can be more easily avoided (i.e. animals), food can be hidden in products without awareness and so a reaction could occur by mistake. This can then result in a significant impact on Quality of Life (QoL) for those with an allergy and their family. Children with peanut allergies reporting more fear of an adverse event and anxiety around managing their condition compared to peers with insulin-dependent diabetes mellitus. In addition, the dietary and social restrictions accompanying the management of food allergy can result in children feeling social isolated or even bullied.

Anxiety is a normal part of human experience as it is an appropriate response to uncertain or unpredictable situations, however when anxiety is excessive it can cause great distress and interfere with daily functioning. In regards to the management of an allergy, some level of anxiety is adaptive as anxious children are less likely to take risks in terms of exposure to the allergen compared to those who are less anxious. However, sometimes the anxiety around a fatal reaction can result in avoidance of social situations, not allowing age appropriate outings or having an excessively restricted diet which could have implications for children's growth and development. The optimal emotional response has been described as 'relaxed readiness' in order to allow for effective food allergy management whilst minimizing more maladaptive aspects of anxiety such as hypervigilance or avoidance.

Research has identified that adolescents and young people are the age group most at risk for fatal anaphylaxis to foods. As well as this, having a food allergy is related to increased risk of anxiety within this age group. Reaching adolescence is usually the development of personal autonomy and independence and for those with food allergies is the time where they take more responsibility for the management of their allergy and the subsequent psychosocial impact. Adolescents report feeling misunderstood by others and speak about the psychological consequences of 'being different'.

Considering the 'relaxed readiness' response, interventions for patients with food allergy should aim to recognise, normalise and support levels of anxiety that can allow for more adaptive coping strategies. Adolescents with more avoidant coping strategies (such as avoiding social events or places where they could be exposed to the allergen) are associated with higher trait anxiety, believed to be linked to years of fear of exposure to their allergen. Coping skills that are developed in adolescent tend to persist into adulthood and those which are more constructive have a more positive impact on wellbeing as well as adherence to medical advice. Therefore, an intervention would be beneficial to target a reduction in maladaptive coping techniques and increase adaptive cognitive behavioural problem-solving approach.

A recent systematic review into the effectiveness of interventions to improve self-management for adolescents with allergic conditions found all interventions that met their criteria to be for asthma, highlighting the need for interventions for those with food allergies. A systematic review into the impact of anaphylaxis and anxiety highlighted the need for Cognitive Behavioural Therapy (CBT) based intervention. CBT has also shown to be effective in supporting children with health conditions in managing distress, increased competence in mastering the challenges of adolescence and improvement in coping skills. Although little is known about CBT for children with food allergies, interventions using CBT for parents of children with food allergies have shown to be effective in reducing levels of worry and anxiety and improving quality of life. In recent research, a single session intervention reduced anxiety in the long term and CBT as a single session intervention has been shown to reduce anxiety in young people with anxiety. As the literature has highlighted feelings of not being understood by peers and feeling different, it may be beneficial to offer adolescents the opportunity to meet others in a similar situation. Group intervention is recommended for adolescents as it can be reassuring that patients concerns are shared and discussions can promote more adaptive ways of coping.

The current study addresses the need highlighted in the literature to provide adolescents who experience increased anxiety due to their food allergy with a CBT based intervention to manage the impact of this. This research will design and provide a one-day group CBT workshop for children ages 11-17 with a food allergy and self-reported anxiety. There will also be an optional interview for those who attended the workshop to discuss how they found it and their experiences of living with a food allergy. The results will contribute to the current literature on how anxiety and food allergy are related as well as the feasibility of delivering a CBT workshop for this client group.

ELIGIBILITY:
Inclusion Criteria:

* Children and Adolescents ages 11-17 years with a food allergy.
* To have reported anxiety or worry in relation to management of food allergy.
* Able to attend the one-day workshop at the University of Surrey to complete the intervention in full (or online alternative).
* Willing and able to comprehend English and provide assent/consent.

Exclusion Criteria:

* Child does not speak English.
* Able and willing to engage and understand the content of the workshop.
* Currently under a mental health team and receiving ongoing psychological input.
* Do not have the capacity to provide informed assent/consent and/or consent not gained from caregivers.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Food Allergy Quality of Life Questionnaire (FAQLQ-CF) - Child Form (8-12 years) or Teenager Form (13-17 years) | Baseline, 1 month & 3 month post follow ups
  Child reported quality of life measure specific to food allergy. The FAQLQ-CF provides a self-report on the child's Health Related Quality of Life and contains 24 items and four domains (Risk of Accidental Exposure, Emotional Impact, Allergen Avoidance and Dietary Restrictions) Items were scored on a seven-point scale ranging from not troubled to extremely troubled. For the child form, in order to improve understanding, the scale was illustrated by drawings of faces ('smileys'), ranging from a smiling face to a sad face. The total FAQLQ score is the sum of all the items divided by the number of items and ranges from 1 (minimal impairment) to 7 (maximal impairment).
Change in Penn State Worry Questionnaire for Children (PSWQ-C) | Baseline, 1 month & 3 month post follow ups
  Child reported worry measure. Respondents are asked to rate how often each item applies to them by choosing from a 4-point Likert scale consisting of never (0), sometimes (1), often (2) and always (3). The scores from each item are summed together to yield a total score that ranges from 0-42, with higher scores reflecting higher levels of worry.

SECONDARY OUTCOMES:
Change in Coping Strategies Inventory (CSI) | Baseline, 1 month & 3 month post follow ups
  Assesses coping thoughts and behaviours in response to a specific stressor (food allergy). After describing a stressful situation, persons taking the CSI are asked to respond to 32 questions in a 5-item Likert format. Respondents indicate for each item the extent to which they performed that particular coping response in dealing with the previously described situation (not at all, a little, somewhat, much, very much). Current scoring practices for the CSI involve giving all items in a particular subscale equalweights. To obtain the raw score for a subscale, simply add the item scores. With the higher score suggesting more use of that strategy.
Change in Adherence to food allergy specific self-care behaviours | Baseline, 1 month & 3 month post follow ups
  Assessment of adherence to food allergy specific self-care behaviours. Questionnaire. Five items. Responses are measured on a 6-point scale (0-5) how much each statement applies to them. Higher the score suggests poorer self-care behaviours.
Change in Food Allergy Quality of Life Questionnaire (FAQLQ-PF)- Parent Form (8-12 years) or Parent Form (13-17 years) | Baseline, 1 month & 3 month post follow ups
  Parent reported survey of child quality of life. The FAQLQ-PF provides a parent report on the child's Health related quality of life and contains 30 items for children aged 0-12 (child form) and 13-17 (teenager form) years. Items are divided into three domains (Emotional Impact, Food Anxiety and Social & Dietary Limitations) and scored in the same way as the FAQLQ-CF.
Intervention Feedback Survey | 3 month post workshop
  Satisfaction and experience with intervention, Client Change Interview Schedule
Change in Goals based outcome measure | Baseline, 1 month & 3 month post follow ups
  Goals from workshop and success at achieving on a scale from 0 (Goal not at all met) to 10 (Goal achieved). The higher the score, the better the outcome.

OTHER OUTCOMES:
Demographics | Baseline
  Food allergy and anxiety characteristics
Feasibility of the intervention in terms of the number interested, recruited and completion of the intervention. | 3 months post workshop
  Number of children invited to the study, number of children interested in participating in the study, number of children meeting eligibility criteria, number of children recruited and participating in the intervention, number of children that completed the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Tallentire, BSc, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

REFERENCES:
- [Background] Loh W, Tang MLK. The Epidemiology of Food Allergy in the Global Context. Int J Environ Res Public Health. 2018 Sep 18;15(9):2043. doi: 10.3390/ijerph15092043. PMID 30231558
- [Background] Muraro A, Werfel T, Hoffmann-Sommergruber K, Roberts G, Beyer K, Bindslev-Jensen C, Cardona V, Dubois A, duToit G, Eigenmann P, Fernandez Rivas M, Halken S, Hickstein L, Host A, Knol E, Lack G, Marchisotto MJ, Niggemann B, Nwaru BI, Papadopoulos NG, Poulsen LK, Santos AF, Skypala I, Schoepfer A, Van Ree R, Venter C, Worm M, Vlieg-Boerstra B, Panesar S, de Silva D, Soares-Weiser K, Sheikh A, Ballmer-Weber BK, Nilsson C, de Jong NW, Akdis CA; EAACI Food Allergy and Anaphylaxis Guidelines Group. EAACI food allergy and anaphylaxis guidelines: diagnosis and management of food allergy. Allergy. 2014 Aug;69(8):1008-25. doi: 10.1111/all.12429. Epub 2014 Jun 9. PMID 24909706
- [Background] Avery NJ, King RM, Knight S, Hourihane JO. Assessment of quality of life in children with peanut allergy. Pediatr Allergy Immunol. 2003 Oct;14(5):378-82. doi: 10.1034/j.1399-3038.2003.00072.x. PMID 14641608
- [Background] Cummings AJ, Knibb RC, Erlewyn-Lajeunesse M, King RM, Roberts G, Lucas JS. Management of nut allergy influences quality of life and anxiety in children and their mothers. Pediatr Allergy Immunol. 2010 Jun;21(4 Pt 1):586-94. doi: 10.1111/j.1399-3038.2009.00975.x. Epub 2010 Jan 14. PMID 20088863
- [Background] Ravid NL, Annunziato RA, Ambrose MA, Chuang K, Mullarkey C, Sicherer SH, Shemesh E, Cox AL. Mental health and quality-of-life concerns related to the burden of food allergy. Psychiatr Clin North Am. 2015 Mar;38(1):77-89. doi: 10.1016/j.psc.2014.11.004. Epub 2014 Dec 20. PMID 25725570
- [Background] Muraro A, Polloni L, Lazzarotto F, Toniolo A, Baldi I, Bonaguro R, Gini G, Masiello M. Comparison of bullying of food-allergic versus healthy schoolchildren in Italy. J Allergy Clin Immunol. 2014 Sep;134(3):749-51. doi: 10.1016/j.jaci.2014.05.043. Epub 2014 Jul 18. No abstract available. PMID 25042742
- [Background] Gross C, Hen R. The developmental origins of anxiety. Nat Rev Neurosci. 2004 Jul;5(7):545-52. doi: 10.1038/nrn1429. No abstract available. PMID 15208696
- [Background] Mandell D, Curtis R, Gold M, Hardie S. Anaphylaxis: how do you live with it? Health Soc Work. 2005 Nov;30(4):325-35. doi: 10.1093/hsw/30.4.325. PMID 16323724
- [Background] Klinnert MD, Robinson JL. Addressing the psychological needs of families of food-allergic children. Curr Allergy Asthma Rep. 2008 May;8(3):195-200. doi: 10.1007/s11882-008-0033-7. PMID 18589837
- [Background] Polloni L, Toniolo A, Lazzarotto F, Baldi I, Foltran F, Gregori D, Muraro A. Nutritional behavior and attitudes in food allergic children and their mothers. Clin Transl Allergy. 2013 Dec 10;3(1):41. doi: 10.1186/2045-7022-3-41. PMID 24325875
- [Background] Walkner M, Warren C, Gupta RS. Quality of Life in Food Allergy Patients and Their Families. Pediatr Clin North Am. 2015 Dec;62(6):1453-61. doi: 10.1016/j.pcl.2015.07.003. Epub 2015 Sep 8. PMID 26456443
- [Background] Turner PJ, Gowland MH, Sharma V, Ierodiakonou D, Harper N, Garcez T, Pumphrey R, Boyle RJ. Increase in anaphylaxis-related hospitalizations but no increase in fatalities: an analysis of United Kingdom national anaphylaxis data, 1992-2012. J Allergy Clin Immunol. 2015 Apr;135(4):956-963.e1. doi: 10.1016/j.jaci.2014.10.021. Epub 2014 Nov 25. PMID 25468198
- [Background] Ferro MA, Van Lieshout RJ, Scott JG, Alati R, Mamun AA, Dingle K. Condition-specific associations of symptoms of depression and anxiety in adolescents and young adults with asthma and food allergy. J Asthma. 2016;53(3):282-8. doi: 10.3109/02770903.2015.1104694. Epub 2016 Jan 21. PMID 26539899
- [Background] MacKenzie H, Roberts G, van Laar D, Dean T. Teenagers' experiences of living with food hypersensitivity: a qualitative study. Pediatr Allergy Immunol. 2010 Jun;21(4 Pt 1):595-602. doi: 10.1111/j.1399-3038.2009.00938.x. Epub 2009 Aug 21. PMID 19702674
- [Background] DunnGalvin A, Gaffney A, Hourihane JO. Developmental pathways in food allergy: a new theoretical framework. Allergy. 2009 Apr;64(4):560-8. doi: 10.1111/j.1398-9995.2008.01862.x. Epub 2009 Jan 9. PMID 19154549
- [Background] Polloni L, Muraro A. Anxiety and food allergy: A review of the last two decades. Clin Exp Allergy. 2020 Apr;50(4):420-441. doi: 10.1111/cea.13548. Epub 2020 Jan 6. PMID 31841239
- [Background] Polloni L, DunnGalvin A, Ferruzza E, Bonaguro R, Lazzarotto F, Toniolo A, Celegato N, Muraro A. Coping strategies, alexithymia and anxiety in young patients with food allergy. Allergy. 2017 Jul;72(7):1054-1060. doi: 10.1111/all.13097. Epub 2017 Jan 11. PMID 27886387
- [Background] Schmidt S, Petersen C, Bullinger M. Coping with chronic disease from the perspective of children and adolescents--a conceptual framework and its implications for participation. Child Care Health Dev. 2003 Jan;29(1):63-75. doi: 10.1046/j.1365-2214.2003.00309.x. PMID 12534568
- [Background] Knibb RC, Alviani C, Garriga-Baraut T, Mortz CG, Vazquez-Ortiz M, Angier E, Blumchen K, Comberiati P, Duca B, DunnGalvin A, Gore C, Hox V, Jensen B, Pite H, Santos AF, Sanchez-Garcia S, Gowland MH, Timmermans F, Roberts G. The effectiveness of interventions to improve self-management for adolescents and young adults with allergic conditions: A systematic review. Allergy. 2020 Aug;75(8):1881-1898. doi: 10.1111/all.14269. PMID 32159856
- [Background] Manassis K. Managing anxiety related to anaphylaxis in childhood: a systematic review. J Allergy (Cairo). 2012;2012:316296. doi: 10.1155/2012/316296. Epub 2011 Oct 5. PMID 22007248
- [Background] Christie D, Wilson C. CBT in paediatric and adolescent health settings: a review of practice-based evidence. Pediatr Rehabil. 2005 Oct-Dec;8(4):241-7. doi: 10.1080/13638490500066622. PMID 16192099
- [Background] Knibb RC. Effectiveness of Cognitive Behaviour Therapy for Mothers of Children with Food Allergy: A Case Series. Healthcare (Basel). 2015 Nov 25;3(4):1194-211. doi: 10.3390/healthcare3041194. PMID 27417820
- [Background] Boyle RJ, Umasunthar T, Smith JG, Hanna H, Procktor A, Phillips K, Pinto C, Gore C, Cox HE, Warner JO, Vickers B, Hodes M. A brief psychological intervention for mothers of children with food allergy can change risk perception and reduce anxiety: Outcomes of a randomized controlled trial. Clin Exp Allergy. 2017 Oct;47(10):1309-1317. doi: 10.1111/cea.12981. Epub 2017 Aug 10. PMID 28710902
- [Background] Sugunasingha N, Jones FW, Jones CJ. Interventions for caregivers of children with food allergy: A systematic review. Pediatr Allergy Immunol. 2020 Oct;31(7):805-812. doi: 10.1111/pai.13255. Epub 2020 Jun 24. PMID 32311157
- [Background] Schleider JL, Weisz JR. Little Treatments, Promising Effects? Meta-Analysis of Single-Session Interventions for Youth Psychiatric Problems. J Am Acad Child Adolesc Psychiatry. 2017 Feb;56(2):107-115. doi: 10.1016/j.jaac.2016.11.007. Epub 2016 Nov 25. PMID 28117056
- [Derived] Jones CJ, Tallentire H, Edgecumbe R, Sherlock G, Hale L. Online, group, low-intensity psychological intervention for adults, children, and parents with food allergy. Ann Allergy Asthma Immunol. 2024 Oct;133(4):453-461. doi: 10.1016/j.anai.2024.07.025. Epub 2024 Jul 26. PMID 39069154